CLINICAL TRIAL: NCT02167620
Title: Metformin in Co-morbid Diabetes or Prediabetes and Serious Mental Illness
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Margaret Hahn, Clinician/Scientist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 007/2014
Record Dates: First submitted 2014-06-17; First posted 2014-06-19 (Estimated); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Diabetes Mellitus, Type 2; Schizophrenia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Schizophrenia | interventions — Metformin; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metformin (Placebo Comparator): Metformin/ placebo will be dispensed on a biweekly basis, and pill counts conducted at each visit.
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator): Metformin/ placebo will be dispensed on a biweekly basis, and pill counts conducted at each visit.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — Metformin will be dispensed on a biweekly basis, and pill counts conducted at each visit.
  Arms: Metformin
Drug: Placebo — Placebo will be dispensed on a biweekly basis, and pill counts conducted at each visit.
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
Schizophrenia is associated with a lifespan shortened by 20 years, due to cardiovascular disease (CVD), with antipsychotic (AP) medications understood to contribute to this risk through associated metabolic side-effects. Metformin, a medication used to treat prediabetes, and diabetes in the general population, holds promise with regard to reduction of AP-related metabolic problems, but has not been directly tested in early episode patients beyond weight loss, nor specifically in patients with diabetes or prediabetes and psychosis. We propose to replicate findings that metformin can reduce weight gain, and dysglycemia uniquely focusing on an early episode population diagnosed with prediabetes or diabetes. To help determine long-term risk/benefit of adjunctive metformin, we propose to look at changes in abdominal and liver fat, two well-established risk factors for CVD. Given links between dysglycemia, obesity with hippocampal volume loss and cognitive dysfunction, we will explore if improvements in metabolic indices are associated in changes in cognition and brain structure.

DETAILED DESCRIPTION:
This is a 16 week, double-blind, randomized pilot study, which proposes to recruit 24 patients with schizophrenia, or schizoaffective disorders (DSM 5), who are overweight or obese (BMI >25) and have prediabetes or type 2 diabetes. Randomization occurs on a 2:1 basis, with 16 patients randomised to metformin, and 8 to placebo. Metfomin/placebo is dispensed monthly. The baseline and /or screening visit includes a physical exam (including anthropometric measures), medical history, fasting blood work (glucose, insulin, HbA1c, lipids, electrolytes, thyroid, liver/kidney function), in addition to a urine drug screen. Women of child-bearing age are given a pregnancy test. Patients who meet inclusion criteria and consent to the study have an oral glucose tolerance test (OGTT), and a baseline abdominal and brain MRI (to respectively assess visceral adiposity, a key risk factor for CV disease, and hippocampal volumes). Anthropometric measures and pill counts are repeated bi-weekly. At week 8, fasting insulin/glucose, HbA1C, and liver function tests are measured. End of study measures (week 16), include the same panel of bloodwork conducted at baseline, as well as a repeat OGTT, and an abdominal and brain MRI. Rountine psychopathology scales, including BPRS, CGI, and CDS will be measured at baseline, and week 16. The Brief Assessment of Cognition in Schizophrenia (BACS) will also be completed at baseline, and study end.

ELIGIBILITY:
Inclusion Criteria:

* Patients within 5 years of diagnosis of schizophrenia, schizoaffective disorder , or bipolar disorder(DSM V), or those younger than 40 years old, regardless of duration of illness
* Co-morbid diagnosis of prediabetes or diabetes (Canadian or American Diabetes Association criteria)

Exclusion Criteria:

* Patients with co-morbid axis, other than nicotine dependence, or cannabis abuse
* Patients with liver, or renal dysfunction,
* Patients with a positive drug urine screen (other than cannabis or nicotine)
* Females with a positive pregnancy test will be excluded.
* Prior trial with metformin, and reported lack of tolerability
* Patients with an A1C > 9.5%, or symptomatic hyperglycemia with metabolic decompensation

Ages: 17 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Actual)
Dates: Start 2014-06; Primary Completion 2018-02 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Improvement in HbA1C derived from Oral glucose tolerance test (Matsuda, index of insulin sensitivity; area under glucose curve; insulin secretion sensitivity index-2 (ISSI-2)) | 3 years
  HbA1c value assessment

SECONDARY OUTCOMES:
Decreases in visceral adiposity | 3 years
  Visceral adiposity assessment via MRI
Decreases in hepatic adiposity | 3 years
  Hepatic adiposity assessment via MRI
Greater than 5% decrease in body weight | 3 years
  Body weight assessment
Improvements in cognition | 3 years
  Cognition assessment
Improvements in hippocampal volume | 3 years
  Cognition assessment

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Hahn, Principal Investigator — Center for Addiction and Mental Health
Locations (1):
- Center for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Agarwal SM, Panda R, Costa-Dookhan KA, MacKenzie NE, Treen QC, Caravaggio F, Hashim E, Leung G, Kirpalani A, Matheson K, Chintoh AF, Kramer CK, Voineskos AN, Graff-Guerrero A, Remington GJ, Hahn MK. Metformin for early comorbid glucose dysregulation and schizophrenia spectrum disorders: a pilot double-blind randomized clinical trial. Transl Psychiatry. 2021 Apr 14;11(1):219. doi: 10.1038/s41398-021-01338-2. PMID 33854039